CLINICAL TRIAL: NCT04601714
Title: Baseline Cohort Study to Assess the Malaria Morbidity in Children Living in Future Malaria Vaccine Candidate Trial Sites
Brief Title: Baseline Cohort Malaria Morbidity Study
Acronym: BLOOMy
Status: Completed | Type: Observational
Sponsor: Groupe de Recherche Action en Sante (Other)
Responsible Party: Principal Investigator, Sodiomon B.Sirima, MD, BA, PhD, Groupe de Recherche Action en Sante
Other Study IDs: Protocol_BLOOMy study
Record Dates: First submitted 2020-10-20; First posted 2020-10-26 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Malaria
Keywords: Malaria; Cohort; Children; Epidemiology
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The BLOOMy study is a longitudinal prospective cohort study of healthy children to assess the incidence of clinical malaria over the main transmission season. Participants will undergo baseline clinical and biological assessments then will receive a curative dose of either artesunate or dihydroartemisinin-piperaquine to clear any existing parasitemia. Clearance of parasites will be confirmed 3 weeks later by Polymerase chain reaction (PCR) and only participants with negative PCR will be definitively enrolled for the longitudinal follow up. Both active and passive case detection will be used to ensure that capture of a high proportion of infections in the cohort is achieved.

Blood samples for immunological assessments will be obtained at Day 0 of each positive blood smear episode before treatment and at Weeks 4 post treatment.

Participants will be followed for a minimum of six months throughout the malaria peak transmission season.

DETAILED DESCRIPTION:
The BLOOMy study has two co-Primary objectives:

* To assess the incidence of clinical malaria meeting the primary case definition in children aged 1.5 to 12 years living in the study area over the main transmission season
* To assess the occurrence of reinfection following the radical cure of existing parasitemia.

The secondary objectives are:

* To assess the incidence of clinical malaria meeting various secondary cases definition in children aged 1.5 to 12 years living in the study area over the main transmission season
* To measure the immune responses (humoral and cell-mediated) to a panel of malaria vaccine candidate antigens
* To assess the molecular force of infection
* To pilot and standardize malaria morbidity assessment in three phase 2 malaria vaccine testing sites.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children aged 1.5 to 12 years
* Residence in the study area or surroundings for the period of the study
* Written informed consent from parents/legally acceptable representatives and an assent for children

Exclusion Criteria:

* Complicated symptomatic malaria (defined according to standard World Health Organization criteria)
* Anaemia (Hb<8g/dL),
* Any (chronic) illness that requires immediate clinical care.
* Family history of sudden death or of congenital or clinical conditions known to prolong QTcB or QTcF interval or e.g. family history of symptomatic cardiac arrhythmias, with clinically relevant bradycardia or severe cardiac disease
* Any treatment which can induce a lengthening of QT interval
* Known history of hypersensitivity or allergic reactions to piperaquine or other aminoquinolones
* Receipt of any blood transfusion or immunoglobulins within 3 months
* Known history of hypersensitivity or allergic reactions to artesunate
* Severe malnutrition (weight-for-height being below -3 standard deviation or less than 70% of median of the World Health Organization (WHO) normalized reference values).
* Weight below 5 kg
* Current or previous participation in malaria vaccine trials
* Current active participation in any trial involving administration of investigational drug.

Ages: 18 Months to 12 Years | Sex: All
Age Groups: Child
Study Population: Healthy children aged 1.5 to 12 years
Sampling Method: Probability Sample
Enrollment: 459 (Actual)
Dates: Start 2020-09-07 (Actual); Primary Completion 2021-09-28 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Number of clinical malaria episodes per child-year at risk meeting the primary case definition | 6 months
  The primary case definition: Positive P. falciparum parasitemia at a density > 0 detected by microscopy associated with measured fever (Axillary temperature ≥37.5°C/Tympanic ≥38°C or Forehead temperature ≥37.5°C using non-contact infrared thermometer))
Time to P. falciparum infection detected by positive thick blood smear within 6 months after the enrolment in African children under natural exposure to P. falciparum by treatment group | 6 months

SECONDARY OUTCOMES:
Number of clinical malaria episodes per child-year at risk meeting the following secondary cases definition | 6 months
  Second Secondary case definition: Measured fever (Axillary temperature ≥37.5°C/Tympanic ≥38°C or Forehead temperature ≥37.5°C using non-contact infrared thermometer) AND parasitemia of >5,000 parasites (p) / μl
Number of new P. falciparum clones acquired over time | 6 months
Immune responses to malaria candidate vaccines in the consortium portfolio | 6 months
  Panel of malaria vaccine candidate's antigens such as PfSPZ CVAC, ME-TRAP, R21 (Pre erythrocytic stage antigens) and PfRH5, NPC-SE36 (Blood stage antigens) will be used to assess antibody responses at day 0 and 28 of confirmed episodes of clinical malaria.

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe de Recherche Action en Santé, Ouagadougou, Burkina Faso

REFERENCES:
- [Result] Tiono AB, Kangoye DT, Rehman AM, Kargougou DG, Kabore Y, Diarra A, Ouedraogo E, Nebie I, Ouedraogo A, Okech B, Milligan P, Sirima SB. Malaria incidence in children in South-West Burkina Faso: comparison of active and passive case detection methods. PLoS One. 2014 Jan 24;9(1):e86936. doi: 10.1371/journal.pone.0086936. eCollection 2014. PMID 24475198
- [Result] Guyant P, Corbel V, Guerin PJ, Lautissier A, Nosten F, Boyer S, Coosemans M, Dondorp AM, Sinou V, Yeung S, White N. Past and new challenges for malaria control and elimination: the role of operational research for innovation in designing interventions. Malar J. 2015 Jul 17;14:279. doi: 10.1186/s12936-015-0802-4. PMID 26185098
- [Derived] Ouedraogo A, Ouattara D, Ouattara SM, Diarra A, Badoum ES, Hema A, Ouedraogo AZ, Hien D, Bougouma EC, Nebie I, Bocquet V, Vaillant M, Tiono AB, Sirima SB. Evaluating artesunate monotherapy and dihydroartemisinin-piperaquine as potential antimalarial options for prevaccination radical cures during future malaria vaccine field efficacy trials. Malar J. 2024 Dec 18;23(1):377. doi: 10.1186/s12936-024-05198-1. PMID 39695728